CLINICAL TRIAL: NCT05335291
Title: Turkish Validity and Reliability Study of Physiotherapist Self-Efficacy Questionnaire
Brief Title: Turkish Validity and Reliability of Physiotherapist Self-Efficacy Questionnaire
Status: Completed | Type: Observational
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, Cigdem Emirza, Research Assistant, Istanbul Bilgi University
Other Study IDs: 20022-40030-32
Record Dates: First submitted 2022-04-06; First posted 2022-04-19 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Physiotherapy; Self Efficacy; Education
Keywords: physiotherapy; self efficacy; clinical practice; validation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group I
  Interventions: Other: Questionnaire study

INTERVENTIONS:
Other: Questionnaire study — The Turkish validity and reliability of the questionnaire will be examined.

SUMMARY:
The aim of this study is to provide Turkish validation and determine the validity of the "Physiotherapist Self-Efficacy Questionnaire".

DETAILED DESCRIPTION:
Self-efficacy is defined as one's belief in one's existing capacity to perform the necessary behavior in a specific situation. "Physiotherapist Self-Efficacy Questionnaire" has been developed to be used in the assessment of self-efficacy for the field of physiotherapy and rehabilitation. In this scale, there are 13 items about how competent the individual feels in clinical assessment, problem solving, planning, and communication related to caseloads.

It has been shown that the scale is a valid and reliable method in cardiorespiratory, musculoskeletal and neurological clinical fields, which are special areas of physiotherapy and rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak, read, understand and write in Turkish
* Physiotherapy and rehabilitation students who have participated in at least one clinical practice
* Physiotherapists working in the clinic

Exclusion Criteria:

* Having cognitive problems

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The physiotherapy and rehabilitation students who have done internship in at least one institution or graduate physiotherapists will be included in the study. Participants will re-answer the Turkish version of Physiotherapist Self-Efficacy Questionnaire within one week. They will also answer the General Self-efficacy Scale.
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-11-03 (Actual)

PRIMARY OUTCOMES:
Turkish version of Physiotherapist Self-Efficacy Questionnaire-cardiorespiratory area | Baseline and after one week
  The questionnaire consists of 13 items. The participants will asked to indicate their confidence to perform the described task (1 = very little confidence; 5 = a lot of confidence). Higher scores are related more confidence self-efficacy.
Turkish version of Physiotherapist Self-Efficacy Questionnaire-musculoskeletal area | Baseline and after one week
  The questionnaire consists of 13 items. The participants will asked to indicate their confidence to perform the described task (1 = very little confidence; 5 = a lot of confidence). Higher scores are related more confidence self-efficacy.
Turkish version of Physiotherapist Self-Efficacy Questionnaire-neurological area | Baseline and after one week
  The questionnaire consists of 13 items. The participants will asked to indicate their confidence to perform the described task (1 = very little confidence; 5 = a lot of confidence). Higher scores are related more confidence self-efficacy.

SECONDARY OUTCOMES:
General Self-Efficacy Scale | Baseline
  This scale consists of 10 items. The answers are in a four-likert form (completely true, somewhat true, moderately accurate, completely wrong).

CONTACTS AND LOCATIONS:
Overall Officials: Aycan Cakmak Reyhan, PT, phD, Principal Investigator — Istanbul Bilgi University; Tugba Kuru Colak, PT, phD, Principal Investigator — Marmara University
Locations (1):
- Istanbul Bilgi University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aypay, A. (2010). The Adaptation Study of General Self-Efficacy (GSE) Scale to Turkish. Inonu University Journal of the Faculty of Education (INUJFE), 11(2).
- [Result] van Lankveld W, Jones A, Brunnekreef JJ, Seeger JPH, Bart Staal J. Assessing physical therapist students' self-efficacy: measurement properties of the Physiotherapist Self-Efficacy (PSE) questionnaire. BMC Med Educ. 2017 Dec 12;17(1):250. doi: 10.1186/s12909-017-1094-x. PMID 29233154